CLINICAL TRIAL: NCT00405106
Title: The Effect of Final Exam Preparation on Anxiety Level, Self-Perception, Ocular Symptoms, Accommodation and Vergence in Myopia
Status: Completed | Type: Observational
Sponsor: Southern California College of Optometry at Marshall B. Ketchum University (Other)
Other Study IDs: 04-4
Record Dates: First submitted 2006-11-27; First posted 2006-11-29 (Estimated); Last update posted 2006-11-29 (Estimated); Status verified 2004-05

CONDITIONS: Myopia
Keywords: stress; anxiety; myopia progression; accommodation; vergence
MeSH Terms: conditions — Myopia; Anxiety Disorders

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
To evaluate the effects of exam preparation on anxiety level, self perception, ocular symptoms and oculomotor responses in myopes

DETAILED DESCRIPTION:
Twenty two first year optometry students were evaluated towards the end of their first academic year on a battery of Oculomotor and Survey tests. This occurred during two sessions, one Low Stress session and one High Stress session. Sessions were separated by one month.

Low Stress Session (LS), No Exams or Minor Exams High Stress Session (HS), Final Exam Preparation week

Battery of Surveys:

Adult Manifest Anxiety Scale for College Students (AMAS-C):

36 items which probe 4 types of anxiety

* Worry/Oversensitivity
* Test Anxiety
* Physiological Anxiety (Somatic responses to anxiety)
* Social Concerns

Self Perception Profile (SPP):

45 items which probe 9 domains

* Scholastic Competence
* Social Acceptance
* Athletic Competence
* Physical Appearance
* Job Competence
* Romantic Appeal
* Behavioral Conduct
* Close Friendship
* Global Self-worth

CI Symptom Survey (CISS-15):

15 items which probe ocular and aesthenopic signs and symptoms

Students also reported Hours of daily near work (NWhrs).

Battery of Oculomotor Tests:

(20/30 ETDRS target used for all) Vergence Tests

* Phorias Near and Far (Neutralized Alternate Cover Test)
* Vergence Ranges Near and Far (Prism Bar)
* Vergence Facility Near and Far (3BI/12BO)
* Near Point of Convergence

Objective Accommodative Tests (SRW-5000autorefractor)

Monocular Accommodative Responses to:

* Near Target (33cm)
* Minus Lens (-3D) while viewing distant (6m) target

Subjective Accommodative Tests:

Monocular Accommodative Responses to:

* Donder's Push Up Amplitude test
* Near Accommodative Facility (+/-2.00, five practice trials)
* Distant Accommodative Facility (plano/-2.00, five practice trials)

ELIGIBILITY:
Inclusion Criteria:

* Any first year optometry student

Exclusion Criteria:

* Previous Refractive surgery, amblyopia, strabismus, RGP wearer

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25
Dates: Start 2005-12; Study Completion 2006-05

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Marran, OD PhD, Principal Investigator — SCCO
Locations (1):
- SCCO, Fullerton, California, United States